CLINICAL TRIAL: NCT06574542
Title: The Diagnostic Yield of Push Enteroscopy in Patients With Passing Melena Without Hematemesis, With Nondiagnostic EGD : A Multicenter Study
Brief Title: The Role of Push Enteroscopy in Patients With Passing Melena With Nondiagnostic EGD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Julajak Limsrivilai, Associate Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Si 484/2019
Record Dates: First submitted 2024-08-25; First posted 2024-08-28 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Melena Due to Gastrointestinal Hemorrhage
Keywords: small bowel bleeding; melena; push enteroscopy; colonoscopy; video capsule endoscopy
MeSH Terms: conditions — Melena | interventions — Double-Balloon Enteroscopy; Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Melena, No Hematemesis, and Nondiagnostic EGD (Experimental): Consecutive patients who presented with melena (defined as black, tarry stools) without hematemesis, in whom EGD did not identify a bleeding source, were included for further investigation
  Interventions: Diagnostic Test: Push enteroscopy (PE); Diagnostic Test: Colonoscopy

INTERVENTIONS:
Diagnostic Test: Push enteroscopy (PE) — All patients enrolled in this study underwent evaluation using push enteroscopy (PE)
Diagnostic Test: Colonoscopy — After push enteroscopy (PE), all patients subsequently underwent a colonoscopy on the same day or the next day. However, if a culprit lesion was identified during PE and the patient was considered at risk for undergoing colonoscopy, the colonoscopy was not performed and was presumed to be negative.

SUMMARY:
Melena is often caused by upper gastrointestinal (GI) bleeding; therefore, esophagogastroduodenoscopy (EGD) is the first preferred diagnostic tool. However, EGD fails to identify the bleeding source in about 25% of cases. Guidelines recommend colonoscopy for the subsequent investigation. However, the diagnostic yield of colonoscopy is reportedly low, varying from 4.76% to 35%. Even when EGD and colonoscopy have been performed, 4% to 15% of bleeding cases remain unexplained, suggesting small bowel origins. While video capsule endoscopy (VCE) is recommended due to its high diagnostic yield and noninvasive nature, its limitations include missing proximal small bowel lesions due to rapid transit and the inability to perform therapeutic interventions. Push enteroscopy (PE) is a straightforward, cost-effective technique with a reported 30% to 50% diagnostic success rate for such obscure GI bleeding. This study aims to evaluate the diagnostic yield of PE compared to colonoscopy in patients presenting with melena, no hematemesis, and negative EGD results.

DETAILED DESCRIPTION:
Melena is generally attributed to bleeding from the upper gastrointestinal (GI) tract, with esophagogastroduodenoscopy (EGD) serving as the primary diagnostic tool. However, EGD fails to detect bleeding sources in approximately 25% of cases, necessitating further investigation into potential mid-to-lower GI bleeding. Current guidelines recommend performing a colonoscopy in patients with melena and a negative EGD result before exploring small bowel sources. The effectiveness of colonoscopy in identifying bleeding sources varies significantly, with large-scale studies indicating a low detection rate of around 4.76%, while smaller studies report higher rates, ranging from 23% to 35%.

Despite thorough evaluations using both EGD and colonoscopy, the cause of overt GI bleeding remains unidentified in 4% to 15% of cases, prompting consideration of small bowel bleeding. Video capsule endoscopy (VCE) is often recommended in this situation due to its high diagnostic yield and noninvasive nature. However, VCE has limitations, such as missing proximal small bowel lesions and the inability to provide therapeutic interventions.

Push enteroscopy (PE) offers an alternative approach for investigating obscure GI bleeding. This straightforward endoscopic technique, which most gastroenterologists can perform without specialized equipment, is cost-effective and diagnostically efficient, with yields ranging from 30% to 50%. Utilizing PE in patients with melena and a negative EGD may help avoid unnecessary procedures like colonoscopy and VCE, ultimately reducing treatment costs.

This study aims to compare the diagnostic effectiveness of push enteroscopy (PE) and colonoscopy in patients presenting with melena, no hematemesis, and negative EGD results.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older.
2. Patients admitted to the hospital for acute gastrointestinal bleeding, presenting with symptoms of melena.
3. Patients who have undergone esophagogastroduodenoscopy (EGD) without identification of the source of gastrointestinal bleeding.
4. Patients who have signed informed consent to participate in the study.

Exclusion Criteria:

1. Patients with symptoms of hematemesis, coffee ground emesis, or detection of blood via a gastric lavage tube.
2. Patients with unstable vital signs before undergoing push enteroscopy.
3. Patients with conditions that contraindicate endoscopy, such as severe asthma or serious cardiac conditions.
4. Patients with a history of bleeding disorders or uncorrectable coagulation abnormalities.
5. Patients who have contraindications to bowel preparation with polyethylene glycol.
6. Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic Yield of Push Enteroscopy | 30 day
  This study aimed to evaluate the diagnostic yield of push enteroscopy in patients presenting with melena, without hematemesis, and with a negative EGD.

SECONDARY OUTCOMES:
Diagnostic Yield of Colonoscopy | 30 day
  This study also aimed to evaluate the diagnostic yield of colonoscopy in the same patient population: those presenting with melena, without hematemesis, and with a negative EGD

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology division, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
We are willing to provide our data to researchers who require it. For example, those who want to do systematic review and meta-analysis.
Supporting Information: Study Protocol
Time Frame: Other researchers can contact us anytime.
Access Criteria: We will provide our protocol and/or data upon request.